CLINICAL TRIAL: NCT01579786
Title: The Treatment of Post Operative Pain in Thyroid Surgery Patients: Perspective Study Acupuncture Versus Pharmacological Treatment
Brief Title: Treatment of Post Operative Pain in Thyroid Surgery Patients: Perspective Study Acupuncture Versus Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Donato Nitti, Ordinary Professor of Surgery, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: university of padova
Record Dates: First submitted 2012-04-03; First posted 2012-04-18 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Post Operative Pain
Keywords: post operative pain; acupuncture
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetaminophen (No Intervention): A group All patients will be treated only with drugs used for this type during the operation and post operative pain controlled with usual acetaminophen drug administration (maximum 3 g/day)
- Acetaminophen and acupuncture (Experimental): B group patients. All patients will receive the standard pharmacological treatment for the operation. Acetaminophen (maximum 3g/day) during all seven days after surgery and patients will be treated with acupuncture the first day after surgery and thirty minutes before the surgical procedure
  Interventions: Procedure: Acetaminophen and acupuncture

INTERVENTIONS:
Procedure: Acetaminophen and acupuncture — All patients will receive acetaminophen (maximum 3g/day) for all seven days after surgery and will receive acupuncture treatment at first day after performing surgery and thirty minutes before operation
  Other Names: Acupuncture
  Arms: Acetaminophen and acupuncture

SUMMARY:
The aim of the study was to evaluate if acupuncture may reduce intraoperative ULTIVA (remifentanil) consumption and post operative pain measured with VAS, italian version Mc Gill Questionnaire Pain and drug consumption (acetaminophen daily consumption).

DETAILED DESCRIPTION:
The aim of the study was to evaluate if acupuncture may reduce intraoperative ULTIVA (remifentanil) consumption and post operative pain measured with VAS, italian version Mc Gill Questionnaire Pain and drug consumption (acetaminophen daily consumption). The study involve patients who underwent thyroid surgery randomised in two groups. A group patients treated with drugs and B group patients treated with drugs and acupuncture.Acupuncture related risk are pain, faint and haematoma.The study will be done in Padova University Hospital (Endocrine Unit.Primary end point will be VAS pain and secondary end points ULTIVA consumption, post operative pain measured with italian version of Mc Gill Questionnaire Pain and acetaminophen daily intake

ELIGIBILITY:
Inclusion Criteria:

* thyroid surgery patients

Exclusion Criteria:

* back severe arthritis
* osteoporosis
* myofascial pain
* rheumatic disease
* fibromyalgia
* systemic cardiovascular and respiratory disease
* hypertension
* drug or alcohol consumption
* mental disease
* cervical trauma
* chronic use of antidepressant
* hypnotic and antihypertensive drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | within the 3rd postoperative day
  Change in intensity of pain from first day after operation and during the seven days after performing surgery

SECONDARY OUTCOMES:
Mc Gill Questionnaire pain | within the 3rd postoperative day
  Change in intensity of pain from the day after operation and during all seven days after performing surgery

OTHER OUTCOMES:
Remifentanil consumption | Intraoperative
Acetaminophen | within 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Professor Nitti, Donato, Study Director — University of Pdova
Locations (1):
- Endocrine Unit, Padova Universitary Hospital, Padua, Padova, Italy